CLINICAL TRIAL: NCT06437249
Title: Children's Dental Anxiety in Relation to Parental Dental Anxiety, Child's Age and Gender and Caries Experience (Cross Sectional Study)
Brief Title: Children's Dental Anxiety in Relation to Parental Dental Anxiety, Child's Age and Gender and Caries Experience
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghadeer Jaafar Ali Jawad, Principal Investigator Ghadeer Jaafar Ali, Cairo University
Other Study IDs: children dental anxiety
Record Dates: First submitted 2024-05-21; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Child Dental Anxiety
Keywords: Parental dental anxiety; Child dental anxiety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determine the relation of of Children's dental anxiety to Parental Dental anxiety, child's age and gender and caries experience will be obtained through written questionnaires (ACDAS) and (CDAS) to the child and parents of children aged 6-8 years old in the clinic.

DETAILED DESCRIPTION:
1. Soft copies of the Abeer children dental anxiety SCALE (ACDAS) Questionnaire and Corah Dental Anxiety Scale (CDAS) Questionnaire.
2. The child's age and gender will be recorded first.
3. Level of anxiety will be recorded by using Heart rate using fingertip pulse oximeter.
4. Dental caries experiences will record by using Dental caries indices (DMF and def)
5. Child dental anxiety will be evaluated from (ACDAS) Questionnaire: The first part is child self-report part, the operator will be answered by ticking the box that corresponds to child dental anxiety, 1 (happy), 2 (Ok), 3 (Scared). The second part about the cognitive part with five questions: three of them answered with (Yes, No) and the other two questions answered with score, 1 (happy), 2 (Ok), 3 (Scared)
6. Parents dental anxiety will be evaluated from (CDAS) Questionnaire. the parents will answer by ticking the answer. The final scores, >9 (Mild anxiety), 9-12 (Moderate anxiety), 13-14 (High anxiety), 15-20 (Sever anxiety).
7. Results will be analyzed by the statistician.
8. Data handling will be supervised by the supervisors.

ELIGIBILITY:
Inclusion Criteria:

1. Children range in age from 6-8 years old.
2. First dental visit.
3. Accompanied by their parents.
4. Both male and female included.

Exclusion Criteria:

1. Children with Physical or mental disabilities.
2. Children who refuse to participate.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Gender: Male and Female.
  2. Age: 6-8 years old
     * in Pediatric Clinic in Pediatric Dentistry and Dental Public Health Department-faculty of Dentistry, Cairo University, Egypt.
     * parents will be interviewed by the examiner and the questionnaire will be filled.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Child dental anxiety | Two months
  Using Abeer children dental anxiety SCALE Questionnaire Score score 1 happy 2 Ok 3 Scared
Level of anxiety | Two months
  record Heart rate number using fingertip pulse oximeter
Caries experience | Two months
  Using dental caries indices ( Decayed Missed Filling and Decayed Exposed to extraction Filling ) in mixed dentition

SECONDARY OUTCOMES:
Parental dental anxiety | Two months
  Using Corah Dental Anxiety Scale Questionnaire Score a = 1, b = 2, c = 3, d = 4, e = 5 Total possible = 20
  * < 9 = mild
  * 9 - 12 = moderate anxiety
  * 13 - 14 = high anxiety
  * 15 - 20 = severe anxiety (or phobia) higher score means worse

CONTACTS AND LOCATIONS:
Overall Officials: Ola Mustafa, professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Almanial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
evaluate the relation between the parental dental anxiety, child age and gender and caries experience on child dental anxiety in a group of Egyptian children.

REFERENCES:
- [Result] Coric A, Banozic A, Klaric M, Vukojevic K, Puljak L. Dental fear and anxiety in older children: an association with parental dental anxiety and effective pain coping strategies. J Pain Res. 2014 Aug 20;7:515-21. doi: 10.2147/JPR.S67692. eCollection 2014. PMID 25187737
- [Result] Corah NL, Gale EN, Illig SJ. Assessment of a dental anxiety scale. J Am Dent Assoc. 1978 Nov;97(5):816-9. doi: 10.14219/jada.archive.1978.0394. PMID 31377
- [Result] Al-Namankany A, Ashley P, Petrie A. The development of a dental anxiety scale with a cognitive component for children and adolescents. Pediatr Dent. 2012 Nov-Dec;34(7):e219-24. PMID 23265158
- [Result] Aditya PVA, Prasad MG, Nagaradhakrishna A, Raju NS, Babu DN. Comparison of effectiveness of three distraction techniques to allay dental anxiety during inferior alveolar nerve block in children: A randomized controlled clinical trial. Heliyon. 2021 Sep 29;7(9):e08092. doi: 10.1016/j.heliyon.2021.e08092. eCollection 2021 Sep. PMID 34632153